CLINICAL TRIAL: NCT06909487
Title: Clinical Characterization of Very and Extremely Preterm Infants Who Received Excess Erythrocyte Transfusions With Respect to HAS 2014 Recommendations
Acronym: CGR EXCESS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2025_843_0069
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Very Preterm and Extremely Preterm Birth; Anemia; Erythrocyte Transfusion; Excess Transfusion
Keywords: Very preterm and extremely preterm birth; Anemia; Erythrocyte transfusion; excess transfusion
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prematurity affects around 60,000 births a year in France. Extremely premature babies are particularly fragile and require multiple erythrocyte transfusions to maintain an effective hemoglobin level for metabolism and continued somatic and neurological development. Many known risk factors, such as multiple blood sampling for biological diagnosis, lead to a more rapid fall in hemoglobin concentration, reducing the amount of oxygen delivered in the tissues. In addition, red blood cell regeneration is very low in premature infants, while the half-life of red blood cells is shorter than in older children and adults. The result is severe anemia. Its main treatment is erythrocyte transfusion. It is associated with biological benefits, but has digestive, ophthalmological, pulmonary, metabolic and neurological side effects. To ensure a good benefit/risk ratio, a commission of the HAS issued recommendations in 2014 for erythrocyte transfusion in premature infants < 32 weeks of amenorrhea in France. Yet many transfusions continue to be performed outside the HAS 2014 criteria. A retrospective monocentric study was carried out in order to understand this situation. Data from premature infants < 31 weeks of amenorrhea (wks) born between July 2022 and July 2024 were collected via computerized hospitalization records (DxCare, Diane and Demserv software). Their transfusion status during the first twenty-eight days of life was analyzed. The HAS decision algorithm was used to identify excess transfusions and develop a patient classification.

ELIGIBILITY:
Inclusion Criteria:

* age : ≤ 28 days of life
* Premature newborn with term of birth < 31 weeks hospitalized in intensive care or neonatology intensive care at CHU Amiens-Picardie (CHU-AP) between July 2022 and July 2024, whether born at CHU-AP maternity unit or transferred secondarily

Exclusion Criteria:

* Newborn with term of birth ≥ 31 weeks and > 28 days of life

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature newborn with term of birth < 31 weeks hospitalized in intensive care or neonatology intensive care at CHU Amiens-Picardie (CHU-AP) between July 2022 and July 2024, whether born at CHU-AP maternity unit or transferred secondarily
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
number preterm infants receiving excess transfusions | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No